CLINICAL TRIAL: NCT02651324
Title: A Prospective, Randomized, Double-Blind, Controlled Trial Evaluating the Efficacy of Ketamine for Improvement in Postoperative Pain Control After Spinal Fusion for Idiopathic Scoliosis
Brief Title: Efficacy of Ketamine for Improvement in Postoperative Pain Control After Spinal Fusion for Idiopathic Scoliosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Albany Medical College (Other)
Responsible Party: Principal Investigator, Farzana Afroze, Anesthesiologist, Albany Medical College
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3497
Record Dates: First submitted 2016-01-06; First posted 2016-01-11 (Estimated); Results first posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Idiopathic Scoliosis; Post-operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Ketamine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Group (Experimental): A ketamine bolus of 0.5mg/kg will be given and then the ketamine infusion of 0.2 mg/kg/hr will be initiated prior to incision. Intra-operative opioids will be at the discretion of the attending anesthesiologist. Postoperative management will include continuation of the study drug as well as a standardized morphine patient-controlled analgesia (PCA) and acetaminophen 15 mg/kg IV every 6 hours. On postoperative day 1, patients are started on ketorolac 0.5 mg/kg up to 15 mg IV q8h. On postoperative day 2 they are transitioned to ibuprofen 10 mg/kg up to 600 mg. The ketamine infusion will continue for 48 hours post operatively at which point the PCA is discontinued and patients are transitioned to oral pain medications (Roxicet or Lortab and Flexeril) as per the current protocol.
  Interventions: Drug: Ketamine
- Placebo (Placebo Comparator): A placebo (saline) will be given in place of ketamine
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ketamine
  Arms: Treatment Group
Other: Placebo
  Other Names: Saline
  Arms: Placebo

SUMMARY:
This study hypothesizes that the addition of a low-dose ketamine infusion to usual post-operative pain management will improve pain control as evidenced by an improvement in post-operative pain scores for patients undergoing spinal fusion for idiopathic scoliosis.

DETAILED DESCRIPTION:
After consenting, patients will be randomized by the pharmacy. In the operating room patients will receive ketamine/placebo 0.5mg/kg bolus prior to the surgical incision, followed by ketamine/placebo 0.2mg/kg continuous infusion up to 48hours. All the patients will also receive 15mg/k IV acetaminophen at the end of the surgery, followed by every 6hr for 48hrs. Rest of the pain regimen will be the usual post-operative pain management for spinal fusion for idiopathic scoliosis, which includes morphine PCA, IV ketorolac from POD 1, and flexaril from POD 1.

All the patients and parents will fill out a survey at 0hr, 24hr and 48hr grading their level of satisfaction with the post-operative pain.

ELIGIBILITY:
Inclusion Criteria:

* ASA I, II, III
* Presenting for spinal fusion for idiopathic scoliosis
* English-speaking and able to give assent

Exclusion Criteria:

* Any contraindication to ketamine
* Previous spinal surgery
* Opioid dependence
* Chronic pain condition
* Significant developmental delay
* Pregnancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Farzana Afroze, MD, Principal Investigator — Albany Medical College
Locations (1):
- Albany Medical Center, Albany, New York, United States

REFERENCES:
- [Background] Bijur PE, Silver W, Gallagher EJ. Reliability of the visual analog scale for measurement of acute pain. Acad Emerg Med. 2001 Dec;8(12):1153-7. doi: 10.1111/j.1553-2712.2001.tb01132.x. PMID 11733293
- [Background] Carstensen M, Moller AM. Adding ketamine to morphine for intravenous patient-controlled analgesia for acute postoperative pain: a qualitative review of randomized trials. Br J Anaesth. 2010 Apr;104(4):401-6. doi: 10.1093/bja/aeq041. Epub 2010 Mar 5. PMID 20207747
- [Background] Cha MH, Eom JH, Lee YS, Kim WY, Park YC, Min SH, Kim JH. Beneficial effects of adding ketamine to intravenous patient-controlled analgesia with fentanyl after the Nuss procedure in pediatric patients. Yonsei Med J. 2012 Mar;53(2):427-32. doi: 10.3349/ymj.2012.53.2.427. PMID 22318834
- [Background] DA Conceicao MJ, Bruggemann DA Conceicao D, Carneiro Leao C. Effect of an intravenous single dose of ketamine on postoperative pain in tonsillectomy patients. Paediatr Anaesth. 2006 Sep;16(9):962-7. doi: 10.1111/j.1460-9592.2006.01893.x. PMID 16918659
- [Background] Green SM, Clark R, Hostetler MA, Cohen M, Carlson D, Rothrock SG. Inadvertent ketamine overdose in children: clinical manifestations and outcome. Ann Emerg Med. 1999 Oct;34(4 Pt 1):492-7. doi: 10.1016/s0196-0644(99)80051-1. PMID 10499950
- [Background] Mathews TJ, Churchhouse AM, Housden T, Dunning J. Does adding ketamine to morphine patient-controlled analgesia safely improve post-thoracotomy pain? Interact Cardiovasc Thorac Surg. 2012 Feb;14(2):194-9. doi: 10.1093/icvts/ivr081. Epub 2011 Nov 28. PMID 22159259
- [Background] Michelet P, Guervilly C, Helaine A, Avaro JP, Blayac D, Gaillat F, Dantin T, Thomas P, Kerbaul F. Adding ketamine to morphine for patient-controlled analgesia after thoracic surgery: influence on morphine consumption, respiratory function, and nocturnal desaturation. Br J Anaesth. 2007 Sep;99(3):396-403. doi: 10.1093/bja/aem168. Epub 2007 Jun 18. PMID 17576969
- [Background] Subramaniam K, Subramaniam B, Steinbrook RA. Ketamine as adjuvant analgesic to opioids: a quantitative and qualitative systematic review. Anesth Analg. 2004 Aug;99(2):482-95, table of contents. doi: 10.1213/01.ANE.0000118109.12855.07. PMID 15271729
- [Background] Tsui BC, Wagner A, Mahood J, Moreau M. Adjunct continuous intravenous ketamine infusion for postoperative pain relief following posterior spinal instrumentation for correction of scoliosis: a case report. Paediatr Anaesth. 2007 Apr;17(4):383-6. doi: 10.1111/j.1460-9592.2006.02134.x. PMID 17359410
- [Background] Yamauchi M, Asano M, Watanabe M, Iwasaki S, Furuse S, Namiki A. Continuous low-dose ketamine improves the analgesic effects of fentanyl patient-controlled analgesia after cervical spine surgery. Anesth Analg. 2008 Sep;107(3):1041-4. doi: 10.1213/ane.0b013e31817f1e4a. PMID 18713926
- [Background] Zakine J, Samarcq D, Lorne E, Moubarak M, Montravers P, Beloucif S, Dupont H. Postoperative ketamine administration decreases morphine consumption in major abdominal surgery: a prospective, randomized, double-blind, controlled study. Anesth Analg. 2008 Jun;106(6):1856-61. doi: 10.1213/ane.0b013e3181732776. PMID 18499623

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 50 participants started but only 49 participants received treatment. Total enrollment would be 49. Recruitment total was 50.
Pre-assignment Details: randomized
Groups:
- Treatment Group: A ketamine bolus of 0.5mg/kg will be given and then the ketamine infusion of 0.2 mg/kg/hr will be initiated prior to incision. Intra-operative opioids will be at the discretion of the attending anesthesiologist. Postoperative management will include continuation of the study drug as well as a standardized morphine patient-controlled analgesia (PCA) and acetaminophen 15 mg/kg IV every 6 hours. On postoperative day 1, patients are started on ketorolac 0.5 mg/kg up to 15 mg IV q8h. On postoperative day 2 they are transitioned to ibuprofen 10 mg/kg up to 600 mg. The ketamine infusion will continue for 48 hours post operatively at which point the PCA is discontinued and patients are transitioned to oral pain medications (Roxicet or Lortab and Flexeril) as per the current protocol.
  Ketamine
- Placebo: A placebo (saline) will be given in place of ketamine
  Placebo
Period: Overall Study
Arm/Group | Treatment Group | Placebo
Started | 25 | 25
Completed | 24 (25 patients were screened and consented, but one patient was excluded due to inability to complete the randomization and received standard treatment of care instead of study drug.) | 25
Not Completed | 1 | 0
Not completed — drug not administered, due dispensing issue | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Group | Placebo | Total
Number analyzed (Participants) | 24 | 25 | 49
Age, Customized [Mean (Standard Deviation); unit: years] — 18 years or less
  years
    mean age | 13.4 (1.72) | 14.7 (2.19) | 14.05 (1.945)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 17 | 39
  Male | 2 | 8 | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants] — NY, USA, Albany medical center Albany, NY
  Participants
    United States | 24 | 25 | 49

OUTCOME MEASURES:

1. Primary Outcome: Patient Satisfaction
Description: All the patients and parent will fill out a survey grading their level of satisfaction with their post-operative pain management. Patient Satisfaction Score from a scale of 1 - 4 was used -
  1. Unsatisfied
  2. Moderately satisfied 3 - Generally satisfied 4 - Very satisfied No other subscales were included.
Time Frame: Through study completion, 48 hours
Population: pediatric patient under 18yrs of age, total Femle 39 and total male 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Group | Placebo
Number analyzed (Participants) | 24 | 20
score on a scale
  patient pain satisfaction scores | 2.75 (0.808) | 2.92 (0.712)
  parent pain satisfaction score | 3.31 (0.805) | 3.13 (0.705)

2. Secondary Outcome: Pain Score
Description: Pain scores will be collected from the nursing sheet. Pain score was measured using "self-rating numeric scale" a scale from 1 to 10, where 1 is minimum pain and 10 is maximum pain.
  No other subscales were done.
Time Frame: Through study completion 48 hours
Population: pediatric patient under 18yrs of age
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Group | Placebo
Number analyzed (Participants) | 24 | 24
score on a scale | 3.17 (1.71) | 3.9 (1.81)

3. Secondary Outcome: Opioid Use
Description: Total Morphine consumption will be collected from Patient Controlled Analgesia (PCA) morphine pump. The secondary outcome measure was total morphine consumption difference in 48hrs.
Time Frame: Through study completion, 48 hours
Population: pediatric patient under the age of 18
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Treatment Group | Placebo
Number analyzed (Participants) | 24 | 25
mg | 0.577 (0.374) | 0.83 (0.466)

4. Secondary Outcome: Length of Stay
Description: Length of hospital stay from surgery to discharge
Time Frame: Through study completion, 48 hours
Population: pediatric patient under age of 18
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Treatment Group | Placebo
Number analyzed (Participants) | 24 | 25
hours | 5.46 (0.721) | 5.52 (0.653)

ADVERSE EVENTS:
Time Frame: we monitored the patients for adverse events for 48hrs after the surgery.
Arm/Group | Treatment Group | Placebo
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/25
Other Adverse Events (participants affected / at risk) | 3/24 | 9/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group (N=24) | Placebo (N=25)
GI symptoms (Gastrointestinal disorders) | 3 (24) | 9 (25) — nausea
cardiac (Cardiac disorders) | 1 (24) | 0 — tachycardia
GI symptoms (Gastrointestinal disorders) | 3 (24) | 3 (25) — Constipation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-07-16): https://cdn.clinicaltrials.gov/large-docs/24/NCT02651324/Prot_SAP_000.pdf